CLINICAL TRIAL: NCT05169502
Title: Identification of Biomarkers for Early Detection of Diabetes Complications by Characterisation of Circulating Endothelial Cells in Human Blood Using Single-cell RNA Sequencing.
Brief Title: Discovering Early Biomarkers in Circulating Endothelial Cells for Diabetes Complications by Single Cell RNA Sequencing
Acronym: CEC4DC
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Principal Investigator, Camilla Blunk Brandt, master of science, phd student at Department of Biomedicine, Aarhus University Hospital
Other Study IDs: 33579; AUFF-NOVA Research Grant (Other Grant/Funding Number: AUFF-E-2019-9-17)
Record Dates: First submitted 2021-11-24; First posted 2021-12-27 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Diabetes; Diabetes Mellitus; Proliferative Diabetic Retinopathy; Diabetic Maculopathy; Circulating Endothelial Cells
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — A 20mL whole blood sample will be collected from each participant, which will be used to isolate the peripheral blood mononuclear cells (PBMCs).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients with diabetes and newly diagnosed proliferative diabetic retinopathy, level 4. (n=10): Inclusion criteria: Type I or II diabetes, habile and age>18 years. Exclusion criteria: Incapacitated or age< 18 years.
  One 20mL blood sample from each patient will be analysed by flow cytometry and single cell RNA sequencing.
  A questionnaire describing the patients general health (gender, age, duration of diabetes, smoking status, blood pressure, BMI and hip/waist ratio) will be made.
- Patients with diabetes and newly diagnosed diabetic maculopathy. (n=10): These patients will be matched 1:1 to the patients with proliferative diabetic retinopathy, regarding gender, age, duration of diabetes, smoking status, and blood pressure.
  One 20mL blood sample from each patient will be analysed by flow cytometry and single cell RNA sequencing.A questionnaire describing the patients general health (gender, age, duration of diabetes, smoking status, blood pressure, BMI and hip/waist ratio) will be made.
- Patients with diabetes without retinopathy, level 0. (n=10): These patients will be matched 1:1 to the patients with proliferative diabetic retinopathy, regarding gender, age, duration of diabetes, smoking status, and blood pressure.
  One 20mL blood sample from each patient will be analysed by flow cytometry and single cell RNA sequencing.A questionnaire describing the patients general health (gender, age, duration of diabetes, smoking status, blood pressure, BMI and hip/waist ratio) will be made.
- Individuals without diabetes and known eye diseases (n=10): These patients will be matched 1:1 to the patients with proliferative diabetic retinopathy, regarding gender, age, smoking status, and blood pressure.
  One 20mL blood sample from each patient will be analysed by flow cytometry and single cell RNA sequencing.A questionnaire describing the patients general health (gender, age, smoking status, blood pressure, BMI and hip/waist ratio) will be made.

SUMMARY:
The purpose of this study is to discover early biomarkers in circulating endothelial cells for diabetes complications, by investigating circulating endothelial cells in blood samples from patients with newly diagnosed proliferative diabetic retinopathy, newly diagnosed maculopathy, patients with diabetes without eye diseases, and individuals without diabetes by single-cell RNA sequencing. The single-cell RNA sequencing analysis will make it possible to fully phenotype diabetes circulating endothelial cells at single-cell level and reveal the first atlas of circulating endothelial cells in humans at both healthy and diabetes conditions.

DETAILED DESCRIPTION:
There is one particular type of ECs, which are circulating in the blood system called circulating endothelial cells (CECs). The common concept of CECs only refers to mature ECs that have been shed from the vascular wall due to impaired vascular functions caused by e.g. diabetes, and hypertension. Mature CECs have thus been proposed as highly valuable targets for diagnosis, treatment, and prognosis of cardiovascular diseases. In healthy individuals, the number of CECs varies from 0 to 7000 per ml of blood and increases significantly in patients with hypertension, diabetes, and cardiovascular diseases. In addition to mature EC, which circulates as CEC. Immature EC, called "circulating endothelial progenitor cells" (cEPC), is reduced in patients with cardiovascular disorders. Based on the highly heterogeneous phenotype of vascular ECs found within and between tissues, it is not surprising that all currently known surface markers for both mature CEC and cEPC are debatable as these studies did not consider ECs heterogeneity. Proliferative diabetic retinopathy (PDR) is a well-defined diabetes complication caused by ECs dysfunction. This study will examine human blood (from healthy individuals, patients with diabetes and PDR or diabetic maculopathy, or without eye disease) and thereby characterize both CEC and cEPC by single-cell RNA sequencing.

This study aims to discover early CEC biomarkers for diabetes complications exemplified with diabetic eye diseases.

Recruitment and scRNA-seq: Blood samples from healthy individuals and patients with diabetes and PDR, diabetic maculopathy, or without eye disease will be recruited from Steno Diabetes Center Aarhus and the Department of Ophthalmology at Aarhus University Hospital. The PBMCs will be freshly isolated from the blood samples followed by CEC enrichment by Fluorescent-Activated Cell Sorting of CD45-CD31+ live cells. Ethical and GDPR approval has been obtained.

ScRNA-seq of CECs: The CD45-CD31+ cells will be processed immediately to single-cell capture and -barcoded cDNA synthesis using the Next GEM Single Cell 3' GEM kit (10x genomics). NGS libraries will be prepared and sequenced using the MGI2000 sequencers from BGI. GenomeDK will be used to supercomputing clusters followed by scRNA-seq analysis and visualization. Integrative multi-model scRNA-seq analyses: Standard scRNA-seq analyses will be carried out to stratify the differential subtypes of CECs and cEPCs and identify ECs subtypes associated with the development of proliferative diabetic retinopathy and diabetic maculopathy. Integrative analysis of scRNA-seq results aims to discover CECs biomarkers which can be used for early diagnosis, prevention and treatment of diabetes complications.

ELIGIBILITY:
Inclusion Criteria:

* Type I or II diabetes
* Habile
* Age> 18 years

Exclusion Criteria:

* Incapacitated
* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients with newly diagnosed proliferative diabetic retinopathy and patients with newly diagnosed diabetic maculopathy will be recruited at department of Ophthalmology at Aarhus University Hospital.
  The healthy individuals and patients with diabetes and without eye diseases will be recruited at Steno Diabetes Center Aarhus, Aarhus University Hospital.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-12 (Actual)

PRIMARY OUTCOMES:
Genome wide expression profile of circulating cells in blood samples from each cohort group | The PBMCs (including circulating endothelial cells) will be freshly isolated from the whole blood sampel, and frozen until all samples are collected (8 months). Afterwards flow cytometry and scRNA-seq analysis will be performed on all samples (2 months).
  Flow cytometry and single-cell RNA sequencing will be used to identify and consolidate potential biomarkers for diabetes complications, by making a genome wide expression profile used to characterise the different phenotypes of circulating cells in each cohort group.

CONTACTS AND LOCATIONS:
Overall Officials: Niels Jessen, Professor, Principal Investigator — Steno Diabetes Center Aarhus, Aarhus Universitet Hospital
Locations (1):
- Steno Diabetes Center Aarhus, Aarhus University Hospiral, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Yes
This project will reveal the first atlas (open acces) of circulating endothelial cells in human at both healthy and diabetes conditions.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will become available in 2024
Access Criteria: Open acces atlas

REFERENCES:
- [Background] Rajendran P, Rengarajan T, Thangavel J, Nishigaki Y, Sakthisekaran D, Sethi G, Nishigaki I. The vascular endothelium and human diseases. Int J Biol Sci. 2013 Nov 9;9(10):1057-69. doi: 10.7150/ijbs.7502. eCollection 2013. PMID 24250251
- [Background] Carmeliet P. Angiogenesis in health and disease. Nat Med. 2003 Jun;9(6):653-60. doi: 10.1038/nm0603-653. PMID 12778163
- [Background] Damani S, Bacconi A, Libiger O, Chourasia AH, Serry R, Gollapudi R, Goldberg R, Rapeport K, Haaser S, Topol S, Knowlton S, Bethel K, Kuhn P, Wood M, Carragher B, Schork NJ, Jiang J, Rao C, Connelly M, Fowler VM, Topol EJ. Characterization of circulating endothelial cells in acute myocardial infarction. Sci Transl Med. 2012 Mar 21;4(126):126ra33. doi: 10.1126/scitranslmed.3003451. PMID 22440735
- [Background] Aird WC. Endothelial cell heterogeneity. Cold Spring Harb Perspect Med. 2012 Jan;2(1):a006429. doi: 10.1101/cshperspect.a006429. PMID 22315715